CLINICAL TRIAL: NCT05016674
Title: Assessment of Cellular and Tissue Characteristics in Lipoaspirates Harvested With the LipoLife System and Stirred by VorFat
Brief Title: Assessment of Cellular and Tissue Characteristics in Lipoaspirates Stirred by VorFat
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no recruitment
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-Lipo-VorFat-21-013
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Laser Assisted Liposuction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laser-assisted liposuction (Experimental): Laser-Assisted Liposuction with the LipoLife system.
  Interventions: Device: LipoLife system

INTERVENTIONS:
Device: LipoLife system — Abdominal Laser-Assisted Liposuction

SUMMARY:
Single-center, prospective, open-label study. The study aims to assess the structure and viability of fat collected during the LipoLife liposuction procedure

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to undergo abdominal w/wo flanks laser-assisted liposuction surgery and are willing to donate the harvested adipose tissue for the study assessment.
2. Between 18 and 70 years of age.
3. Estimated fat harvesting of at least 300 milliliters.
4. Provided written Informed Consent.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the course of study.
2. Current smoker.
3. Presence of known malignancy.
4. Active infection in the treatment area.
5. History of autoimmune disorder (e.g., Systemic Lupus Erythematosus [SLE]).
6. History of connective, metabolic, or atrophic skin disease.
7. History of keloid scarring.
8. Chronic use (>7 consecutive days) of anticoagulants (such as aspirin) or NSAIDs within 15 days before enrollment.
9. Subjects with immune system diseases.
10. Any other reason that in the opinion of the investigator, prevents the subject from participating in the study or compromises the subject safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Average adipose cell cluster size | 6 months
  Assessment of adipose cell cluster size by microscope

CONTACTS AND LOCATIONS:
Overall Officials: William Jason Martin, MD, Principal Investigator — Jason Martin, M.D.
Locations (1):
- William Jason Martin, MD, Denver, Colorado, United States